CLINICAL TRIAL: NCT06940960
Title: An Early Exploratory Clinical Study on the Safety, Tolerability and Preliminary Efficacy of JY231 Injection in the Treatment of Relapsed or Refractory B-Cell Lymphoma/Leukemia
Brief Title: JY231(JY231) Injection for the Treatment of Relapsed/Refractory B Cell Lymphoma/ Leukemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Guangdong Medical University (Other)
Responsible Party: Principal Investigator, Jinqi Huang, associate chief physician, Affiliated Hospital of Guangdong Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JY-CT-24-009
Record Dates: First submitted 2025-03-27; First posted 2025-04-23 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: B Acute Lymphoblastic Leukemia; B-Non Hodgkin Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- A single-center, open, single arm study (Experimental): JY231 Injection for the Treatment of relapsed/refractory B cell lymphoma/ leukemia Subjects who meet the Inclusion Criteria will receive intravenous JY231. JY231 infusion will produce in vivo CAR-T cells in the body.
  Interventions: Drug: JY231 Injection

INTERVENTIONS:
Drug: JY231 Injection — This is an open-label, single-arm study to evaluate the efficacy and safety of in vivo Chimeric Antigen Receptor T-Cell (CAR-T) therapy in patients with relapsed refractory B-cell lymphoma/ leukemia. Upon enrollment, subjects will receive an intravenous infusion of the JY231 preparation. Following the infusion, subjects will be hospitalized for one month for observation, and subjects will be evaluated for safety and efficacy. Subjects will be followed for up to 2 years to determine if the disease is under control.

SUMMARY:
This study is an investigator-initiated single center, single arm clinical study with a target population of patients with relapsed or refractory B cell lymphoma / leukemia. It is an early exploratory clinical study of the safety, tolerability and initial efficacy of JY231 injection in the treatment of relapsed or refractory B cell lymphoma / leukemia.

DETAILED DESCRIPTION:
This open-label, single-arm study is designed to evaluate the efficacy and safety of in vivo CAR-T cell therapy in patients with relapsed/refractory B cell lymphoma/leukaemia. Upon enrolment, leukapheresis will be performed and patients will receive 3-5 days of fludarabine and cyclophosphamide lymphodepleting therapy followed by an intravenous infusion of the JY231 preparation. Following the infusion, subjects will be evaluated for safety and efficacy for up to 24 months to determine if the disease is under control.

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily sign informed consent and are willing and able to comply with all trial requirements;
2. Age is 12-75 years old and gender is not limited;
3. Malignancy cells in bone marrow or peripheral blood are Cluster of Differentiation 19 - positive(CD19+) detected by flow cytometric analysis;
4. Meet the clinical criteria for relapsed or refractory B-cell lymphoma, including: indolent lymphoma (iNHL), such as follicular lymphoma (FL) and marginal zone lymphoma (MZL); aggressive B-cell lymphoma, like diffuse large B-cell lymphoma (DLBCL), primary mediastinal large B-cell lymphoma (PMBCL), transformed follicular lymphoma (TFL), and T-rich lymphocyte-bearing large B-cell lymphoma (TCRBCL), or have a diagnosis of acute B-lymphocytic leukemia (B-ALL) and meet one of the following conditions:

   1. Refractory B-ALL: those who did not achieve complete remission after 2 courses of standard induction regimen chemotherapy, or those who did not achieve complete remission after first-line or multi-line salvage chemotherapy;
   2. Relapsed B-ALL: relapse within 12 months after first remission, or relapse after first-line / multi-line salvage chemotherapy;
   3. Relapse after autologous or allogeneic hematopoietic stem cell transplantation;
   4. In addition, patients with Philadelphia chromosome positive (Ph +) should be relapsed after at least two tyrosine kinase inhibitors (TKI) treatment, or they could not tolerate TKI therapy, or have a t315i mutation, resistant to TKI drugs.
5. Morphological examination of bone marrow cells showed the proportion of primitive and naive lymphocytes was> 5%;
6. No Hematopoietic Stem Cell Transplantation(HSCT) within 6 months before enrollment;
7. At least one measurable lesion was imaging for relapsed or refractory B cell lymphoma, long diameter of> 15mm, or extranodal lesion of> 10mm, along with a positive Positron Emission Tomography - Computed Tomography(PET-CT) examination.
8. More than 12 weeks of expected survival period
9. Baseline Eastern Cooperative Oncology Group(ECOG) score was 0-1;
10. Adequate organ function (criteria regarding liver and kidney function can be moderately relaxed):

    1. Glutamic aminotransferase (ALT) ≤3 times upper limit of normal (ULN);
    2. Grass aminotransferase (AST) ≤3 times ULN;
    3. Total bilirubin ≤1.5 times ULN;
    4. Serum creatinine ≤ 1.5 times ULN, or creatinine clearance ≥ 60 mL/min;
    5. Indoor oxygen saturation ≥ 92%;
    6. Left ventricular ejection fraction (LVEF)≥55%, echocardiography confirmed no pericardial effusion and no clinically significant ECG findings;
    7. There is no clinically significant pleural effusion;
11. Adequate bone marrow reserve without transfusion, defined as:

    1. Absolute neutrophil count (ANC)>1.000 / mm3;
    2. Absolute lymphocyte count (ALC)≥ 300 / mm3;
    3. Platelet≥50.000/mm3;
    4. Hemoglobin>8.0 g/dl;
12. Subjects using the following drugs need to meet the following conditions:

    1. Steroids: The therapeutic dose of steroids must be stopped 72 hours before JY231 infusion. However, physiological alternative doses of steroids are allowed;
    2. Immunosuppression: Any immunosuppressive drug must be stopped at ≥4 weeks prior to enrollment;
    3. Antiproliferative therapy other than lymphodepletion chemotherapy within two weeks of infusion;
    4. Cluster of Differentiation 20(CD20) antibody-related therapy must be stopped within 4 weeks before infusion or 5 half-lives after the CD20 antibody;
    5. CNS disease prophylaxis must be stopped 1 week before JY231 infusion (e. g. intrathecal methotrexate).
13. Reproductive men, sexual partners ensure effective contraception; fertile women, adopted effective contraception and agreed to use contraception throughout the study period.

Exclusion Criteria:

1. Subjects with active cerebrospinal fluid malignant cells or brain metastases, or subjects with active central nervous system (CNS) lymphoma, or CNS leukaemia;
2. Subjects with a history of active CNS disease, such as seizures, cerebrovascular ischemia / hemorrhage, dementia, cerebellar disease, or any autoimmune disease associated with CNS involvement;
3. Subjects who have received other study drugs within 30 days before screening, or are still in the washout period;
4. Patients who have previously received any anti-CD19 / anti-Cluster of Differentiation 3(CD3) therapy or any other anti-CD19 therapy (except for those with normal T cell numbers and function and with CD19-positive tumors);
5. Patients who have been previously treated with any gene therapy product, including Chimeric Antigen Receptor T(CAR-T) therapy (except patients who do not have CAR-T cells in vivo and have normal T cell number and function and are with CD19 positive tumors);
6. Subjects with radiation therapy within 2 weeks prior to the infusion;
7. Subjects with active hepatitis B (defined as Hepatitis B Virus(HBV) DNA test value> 500 IU / mL) or hepatitis C (HCV RNA positive); subjects with HIV positive or treponema pallidum positive;
8. Subjects with uncontrolled acute life-threatening bacterial, viral, or fungal infection (e. g. positive blood culture 72 hours before infusion);
9. Subjects with unstable angina pectoris and / or myocardial infarction within the 6 months prior to screening;
10. Subjects with concurrent or previously diagnosed with other malignancies, except for the patients under following conditions:

    1. Well treated basal cells, papillary thyroid carcinoma, squamous cell carcinoma (adequate wound healing is required before enrollment into this study);
    2. Carcinoma in situ of cervical cancer or breast cancer, after curative treatment, showed no signs of recurrence for at least 3 years before the study;
    3. The primary malignancy has been completely removed and is in complete remission for 5 years.
11. Arrhythmic subjects without medical management control;
12. Subjects receiving oral anticoagulation within 1 week before JY231 injection infusion;
13. Having active neurological autoimmune or inflammatory conditions (such as Guillain-Barre syndrome, amyotrophic lateral sclerosis);
14. Female subjects in pregnant or lactating, or women with planned pregnancy within 2 years after JY231 infusion or male partner with planned pregnancy within 2 years after JY231 infusion;
15. Subjects with taboo study procedures or other medical conditions that may put them at unacceptable risk according to the investigator's judgment and / or clinical criteria.
16. Other conditions that the investigator believes that the subjects should not be enrolled in this clinical trial, such as poor compliance.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events(AE) after infusion | Day 28、Month 2、Month 3、Month 6、Month 12、Month 18、Month 24
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included
Maximal Tolerated Dose(MTD) | Up to 28 days after infusion
  MTD will be determined based on Dose-Limiting Toxicity(DLTs) observed during the first 28 days of study treatment.

SECONDARY OUTCOMES:
Objective Response Rate | Up to 3 months after infusion
  Objective Response Rate(ORR) is defined as the proportion of subjects achieving complete remission(CR) and partial response(PR)

CONTACTS AND LOCATIONS:
Overall Officials: Jinqi Huang, PhD, Principal Investigator — Guangzhou First People's Hospital
Locations (1):
- Affiliated Hospital of Guangdong Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No